CLINICAL TRIAL: NCT00005391
Title: Pediatric Cardiomyopathy Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4297; R01HL053392 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cardiomyopathies

SUMMARY:
To establish and maintain a national registry of children with different forms of cardiomyopathy.

DETAILED DESCRIPTION:
BACKGROUND:

Children with cardiomyopathy represent the most dismal outcome of any group of diseases followed by pediatric cardiologists, with up to 40 percent of infants and children with symptomatic cardiomyopathy failing medical or surgical management in the first year following diagnosis. For 57 percent of children with cardiomyopathy, no etiology is known. Although pediatric cardiomyopathy is common, there is considerable variation in its causes. Therefore, for any specific etiology, no center of pediatric cardiology sees a sufficient number of patients to make major advances in understanding this group of diseases. The registry was developed to collect and organize all relevant data on the condition. Data accrued by and reported by the registry should lead to increased awareness and knowledge of pediatric cardiomyopathy and its causes, as well as the development of new diagnostic and therapeutic approaches.

DESIGN NARRATIVE:

The registry consists of a prospective, population-based cohort of patients in New England and the Central Southwestern United States and a retrospective cohort of patients diagnosed between 1991 and 1996. Annual follow-up data are collected on all patients.

Specific hypotheses are that l) during the period of the registry, the percentage of cases that are diagnosed as idiopathic will decrease (i.e., etiologies will be found) and 2) at the time of diagnosis of cardiomyopathy, factors such as gender, ethnicity, age, type of cardiomyopathy, and presence or absence of a syndrome can help predict outcomes. Definition of entry and exclusion criteria, clinical quality assurance, and accrual and retention of participating clinical centers are largely under the direction of the University of Rochester in Rochester, New York and Baylor College of Medicine. Virtually all pediatric cardiology centers in the United States, Puerto Rico, and Canada have expressed their willingness to send patient information to such a registry.

The study was continued through May, 2010 to to investigate the natural history of cardiomyopathy and transplantation, establish a longitudinal cohort for investigating the functional status of children with cardiomyopathy, and conduct viral and genetic testing to assess associations of genetic and viral markers of cardiomyopathy with clinical and functional outcomes. There are three specific aims. The first expands on the natural history of cardiomyopathy and transplantation by integrating the Pediatric Cardiomyopathy Registry (PCMR) and the Pediatric Heart Transplant Study databases in order to examine whether and how cardiac transplantation modifies the clinical course of cardiomyopathy in children. The second specific aim focuses on the functional status of pediatric cardiomyopathy patients. The study will establish the longitudinal course of functional status in children with cardiomyopathy, and analyze the relationship to clinical events and outcomes. This will be accomplished by assessment of the functional status of pediatric cardiomyopathy patients, including the subset of children undergoing heart transplantation, by continuation of the current PCMR Functional Status Substudy and extension of the study to children in the post-transplant-period period. The third specific aim relates to viral and genetic testing and will investigate how genetic and viral markers of cardiomyopathy are associated with clinical and functional outcomes. Cardiac tissue and blood samples will be collected from 300 children with cardiomyopathy for viral genome and genetic screening 9G4.5 gene) using the Pediatric Cardiomyopathy Repository, and the results will be correlated to clinical outcome.

ELIGIBILITY:
No eligibility criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1995-09; Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lipshultz — University of Miami

REFERENCES:
- [Background] Grenier MA, Osganian SK, Cox GF, Towbin JA, Colan SD, Lurie PR, Sleeper LA, Orav EJ, Lipshultz SE. Design and implementation of the North American Pediatric Cardiomyopathy Registry. Am Heart J. 2000 Feb;139(2 Pt 3):S86-95. doi: 10.1067/mhj.2000.103933. PMID 10650321
- [Background] Bowles KR, Zintz C, Abraham SE, Brandon L, Bowles NE, Towbin JA. Genomic characterization of the human peptidyl-prolyl-cis-trans-isomerase, mitochondrial precursor gene: assessment of its role in familial dilated cardiomyopathy. Hum Genet. 1999 Dec;105(6):582-6. doi: 10.1007/s004399900173. PMID 10647893
- [Background] Lipshultz SE, Fisher SD, Lai WW, Miller TL. Cardiovascular monitoring and therapy for HIV-infected patients. Ann N Y Acad Sci. 2001 Nov;946:236-73. doi: 10.1111/j.1749-6632.2001.tb03916.x. PMID 11762991
- [Background] Lipshultz SE, Sleeper LA, Towbin JA, Lowe AM, Orav EJ, Cox GF, Lurie PR, McCoy KL, McDonald MA, Messere JE, Colan SD. The incidence of pediatric cardiomyopathy in two regions of the United States. N Engl J Med. 2003 Apr 24;348(17):1647-55. doi: 10.1056/NEJMoa021715. PMID 12711739
- [Background] Benun J, Fisher SD, Orav EJ, Schwartz ML, Exil V, Messere C, Lipshultz SE. Cardiac management by pediatricians versus pediatric cardiologists in an inpatient academic center. Am Heart J. 2003 Mar;145(3):424-9. doi: 10.1067/mhj.2003.173. PMID 12660664
- [Background] Lipshultz SE, Lipsitz SR, Sallan SE, Simbre VC 2nd, Shaikh SL, Mone SM, Gelber RD, Colan SD. Long-term enalapril therapy for left ventricular dysfunction in doxorubicin-treated survivors of childhood cancer. J Clin Oncol. 2002 Dec 1;20(23):4517-22. doi: 10.1200/JCO.2002.12.102. PMID 12454107
- [Background] Bergmann SR, Herrero P, Sciacca R, Hartman JJ, Rubin PJ, Hickey KT, Epstein S, Kelly DP. Characterization of altered myocardial fatty acid metabolism in patients with inherited cardiomyopathy. J Inherit Metab Dis. 2001 Nov;24(6):657-74. doi: 10.1023/a:1012711009687. PMID 11768585
- [Background] Lipshultz SE, Rifai N, Dalton VM, Levy DE, Silverman LB, Lipsitz SR, Colan SD, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Gelber RD, Sallan SE. The effect of dexrazoxane on myocardial injury in doxorubicin-treated children with acute lymphoblastic leukemia. N Engl J Med. 2004 Jul 8;351(2):145-53. doi: 10.1056/NEJMoa035153. PMID 15247354
- [Background] Mone SM, Gillman MW, Miller TL, Herman EH, Lipshultz SE. Effects of environmental exposures on the cardiovascular system: prenatal period through adolescence. Pediatrics. 2004 Apr;113(4 Suppl):1058-69. PMID 15060200
- [Background] Adams MJ, Lipsitz SR, Colan SD, Tarbell NJ, Treves ST, Diller L, Greenbaum N, Mauch P, Lipshultz SE. Cardiovascular status in long-term survivors of Hodgkin's disease treated with chest radiotherapy. J Clin Oncol. 2004 Aug 1;22(15):3139-48. doi: 10.1200/JCO.2004.09.109. PMID 15284266
- [Background] Lipshultz SE, Vlach SA, Lipsitz SR, Sallan SE, Schwartz ML, Colan SD. Cardiac changes associated with growth hormone therapy among children treated with anthracyclines. Pediatrics. 2005 Jun;115(6):1613-22. doi: 10.1542/peds.2004-1004. PMID 15930224
- [Background] Lipshultz SE, Lipsitz SR, Sallan SE, Dalton VM, Mone SM, Gelber RD, Colan SD. Chronic progressive cardiac dysfunction years after doxorubicin therapy for childhood acute lymphoblastic leukemia. J Clin Oncol. 2005 Apr 20;23(12):2629-36. doi: 10.1200/JCO.2005.12.121. PMID 15837978
- [Derived] Schmitt W, Diedrich C, Hamza TH, Meyer M, Eissing T, Breitenstein S, Rossano JW, Lipshultz SE. NT-proBNP for Predicting All-Cause Death and Heart Transplant in Children and Adults with Heart Failure. Pediatr Cardiol. 2025 Mar;46(3):694-703. doi: 10.1007/s00246-024-03489-7. Epub 2024 May 9. PMID 38722325
- [Derived] Kantor PF, Shi L, Colan SD, Orav EJ, Wilkinson JD, Hamza TH, Webber SA, Canter CE, Towbin JA, Everitt MD, Pahl E, Ware SM, Rusconi PG, Lamour JM, Jefferies JL, Addonizio LJ, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators*. Progressive Left Ventricular Remodeling for Predicting Mortality in Children With Dilated Cardiomyopathy: The Pediatric Cardiomyopathy Registry. J Am Heart Assoc. 2024 Jan 16;13(2):e022557. doi: 10.1161/JAHA.121.022557. Epub 2024 Jan 12. PMID 38214257
- [Derived] Castleberry CD, Jefferies JL, Shi L, Wilkinson JD, Towbin JA, Harrison RW, Rossano JW, Pahl E, Lee TM, Addonizio LJ, Everitt MD, Godown J, Mahgerefteh J, Rusconi P, Canter CE, Colan SD, Kantor PF, Razoky H, Lipshultz SE, Miller TL. No Obesity Paradox in Pediatric Patients With Dilated Cardiomyopathy. JACC Heart Fail. 2018 Mar;6(3):222-230. doi: 10.1016/j.jchf.2017.11.015. Epub 2018 Feb 7. PMID 29428438
- [Derived] Singh RK, Canter CE, Shi L, Colan SD, Dodd DA, Everitt MD, Hsu DT, Jefferies JL, Kantor PF, Pahl E, Rossano JW, Towbin JA, Wilkinson JD, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators. Survival Without Cardiac Transplantation Among Children With Dilated Cardiomyopathy. J Am Coll Cardiol. 2017 Nov 28;70(21):2663-2673. doi: 10.1016/j.jacc.2017.09.1089. PMID 29169474
- [Derived] Rusconi P, Wilkinson JD, Sleeper LA, Lu M, Cox GF, Towbin JA, Colan SD, Webber SA, Canter CE, Ware SM, Hsu DT, Chung WK, Jefferies JL, Cordero C, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators. Differences in Presentation and Outcomes Between Children With Familial Dilated Cardiomyopathy and Children With Idiopathic Dilated Cardiomyopathy: A Report From the Pediatric Cardiomyopathy Registry Study Group. Circ Heart Fail. 2017 Feb;10(2):e002637. doi: 10.1161/CIRCHEARTFAILURE.115.002637. PMID 28193717
- [Derived] Sleeper LA, Towbin JA, Colan SD, Hsu D, Orav EJ, Lemler MS, Clunie S, Messere J, Fountain D, Miller TL, Wilkinson JD, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators. Health-Related Quality of Life and Functional Status Are Associated with Cardiac Status and Clinical Outcome in Children with Cardiomyopathy. J Pediatr. 2016 Mar;170:173-80.e1-4. doi: 10.1016/j.jpeds.2015.10.004. Epub 2015 Dec 22. PMID 26725459
- [Derived] Everitt MD, Sleeper LA, Lu M, Canter CE, Pahl E, Wilkinson JD, Addonizio LJ, Towbin JA, Rossano J, Singh RK, Lamour J, Webber SA, Colan SD, Margossian R, Kantor PF, Jefferies JL, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators. Recovery of echocardiographic function in children with idiopathic dilated cardiomyopathy: results from the pediatric cardiomyopathy registry. J Am Coll Cardiol. 2014 Apr 15;63(14):1405-13. doi: 10.1016/j.jacc.2013.11.059. Epub 2014 Feb 19. PMID 24561146
- [Derived] Webber SA, Lipshultz SE, Sleeper LA, Lu M, Wilkinson JD, Addonizio LJ, Canter CE, Colan SD, Everitt MD, Jefferies JL, Kantor PF, Lamour JM, Margossian R, Pahl E, Rusconi PG, Towbin JA; Pediatric Cardiomyopathy Registry Investigators. Outcomes of restrictive cardiomyopathy in childhood and the influence of phenotype: a report from the Pediatric Cardiomyopathy Registry. Circulation. 2012 Sep 4;126(10):1237-44. doi: 10.1161/CIRCULATIONAHA.112.104638. Epub 2012 Jul 27. PMID 22843787
- [Derived] Pahl E, Sleeper LA, Canter CE, Hsu DT, Lu M, Webber SA, Colan SD, Kantor PF, Everitt MD, Towbin JA, Jefferies JL, Kaufman BD, Wilkinson JD, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators. Incidence of and risk factors for sudden cardiac death in children with dilated cardiomyopathy: a report from the Pediatric Cardiomyopathy Registry. J Am Coll Cardiol. 2012 Feb 7;59(6):607-15. doi: 10.1016/j.jacc.2011.10.878. PMID 22300696
- [Derived] Foerster SR, Canter CE, Cinar A, Sleeper LA, Webber SA, Pahl E, Kantor PF, Alvarez JA, Colan SD, Jefferies JL, Lamour JM, Margossian R, Messere JE, Rusconi PG, Shaddy RE, Towbin JA, Wilkinson JD, Lipshultz SE. Ventricular remodeling and survival are more favorable for myocarditis than for idiopathic dilated cardiomyopathy in childhood: an outcomes study from the Pediatric Cardiomyopathy Registry. Circ Heart Fail. 2010 Nov;3(6):689-97. doi: 10.1161/CIRCHEARTFAILURE.109.902833. Epub 2010 Sep 10. PMID 20833772